CLINICAL TRIAL: NCT02090400
Title: Multi-centre, Randomized, Open Label Trial to Evaluate the Effects of Switching to Bazedoxifene in Comparison With Switching to Calcium and Vitamin D in Postmenopausal Women Previously Treated With Bisphosphonates
Brief Title: Switching From Oral Bisphosphonates to Bazedoxifene to Evaluate Effects on Bone Mineral Density in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Palacios (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IP-2012-01; 2012-003131-28 (EudraCT Number)
Record Dates: First submitted 2014-03-11; First posted 2014-03-18 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Women; Osteoporosis, Postmenopausal; Bazedoxifene; BMD
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — bazedoxifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bazedoxifene & Calcium/Vit D (Other): Bazedoxifene 20mg oral once a day and calcium 500mg and 400 IU vitamin D (OSTINE)
  Interventions: Drug: Bazedoxifene; Drug: Calcium/Vit D
- Calcium/Vit D (Other): Calcium 500mg and 400 IU vitamin D (OSTINE )daily.
  Interventions: Drug: Calcium/Vit D

INTERVENTIONS:
Drug: Bazedoxifene — 20 mg Oral daily for 12 months
  Other Names: Conbriza
  Arms: Bazedoxifene & Calcium/Vit D
Drug: Calcium/Vit D — Calcium 500 mg / 400 IU Vit D
  Other Names: Ostine

SUMMARY:
The aim of this study is see the changes in bone mineral density after discontinuation or stop the use of bisphosphonates and make the switch to bazedoxifene).

DETAILED DESCRIPTION:
The primary hypothesis is: "Comparing to control group (Calcium+VitD), Bazedoxifene group (20mg daily+ calcium+VitD) is efficient in reducing BMD in spine at 12 months of treatment. in postmenopausal women switching from daily, weekly or monthly bisphosphonates therapy. It is a non-inferiority study of Bazedoxifene compared to biphosphonates, being each patient its own control from the baseline. It is a superiority study of Bazedoxifene compared to Calcium+VitD.

Taking into account the difference in the percentage change observed in the total BMD of the spine during 12 months in those patients treated with Bazedoxifene+Ca+VitD at least 110 patients should be included, 55 in each arm of treatment.

This simple size is going to allow us to detect the differences in the percentage change observed in the total BMD of the spine during 12 months between the two treatment arms, being the same or over 0.25%, with a significance level of 95%, an 80% power. It is estimated a standard deviation of 0.5%, and a 10% lost follow-up rate.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory postmenopausal women 55 years or older at screening
* Have received daily, weekly or monthly oral bisphosphonates at least for 3 years and treatment change is indicated (not responses to bisphosphonates, for bad tolerability or for the potential risk of side effects in a long term treatment with bisphosphonates-indicated by Federal Drug Administration, European Medicines Agency.
* Subjects has stop bisphosphonates therapy no more than one month before screening visit for subjects in daily or weekly bisphosphonates
* Subjects has stop bisphosphonates therapy no more than two months before screening visit for subjects in monthly bisphosphonates
* Screening T-score at the lumbar spine ≤ -2.0 to -4.0 by Dual X ray Absorptiometry (DXA) scan
* At least 2 lumbar vertebrae must be evaluable by DXA
* Al least one hip must be evaluable by DXA (for secondary objectives)

Exclusion Criteria:

* Any disorder that compromises the ability of the subject to give written informed consent and/or to comply with study procedures
* Current use of medication prescribed for osteoporosis other than oral bisphosphonates
* Subjects who had received intravenous bisphosphonates or fluoride (except for dental treatment)
* Subjects who had received any Selective Estrogens Receptor Modulator (SERM), anabolic steroids, systemic hormone replacement, calcitonin or calcitriol within 3 months.
* Subjects who had received strontium ranelate, parathyroid hormone (PTH) or PTH derivates within 1 year.
* Hyper or hypothyroidism, current hyper or hypoparathyroidism
* History of Venous Thromboembolism Event (VTE)
* Significantly impaired renal function as determined by estimated Glomerular Filtration Rate less 35 mL/min
* Hyper or hypocalcemia
* Vitamin D deficiency (serum 25 (OH) vit D level < 20 ng/mL (< 50nmol/L)
* Any condition that could result in impaired calcium metabolism or metabolic bone disease that could interfere with interpretation findings

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Lumbar Spine Bone Mineral Density (BMD) | 12 months
  To evaluate the change in Lumbar Spine Bone Mineral Density (BMD)

SECONDARY OUTCOMES:
Bone Turnover Markers (BTM´s) carboxy-terminal collagen crosslinks (CTX) and 1 procollagen N-terminal (P1NP) | 6 and 12 months from baseline
  To evaluate the effects of switching to Bazedoxifene 20mg in comparison with switching to calcium 500mg and 400 International Units (IU) vitamin D (OSTINE) daily on BTM's CTX and P1NP
BMD at the femoral neck | 6 and 12 months from baseline
  To evaluate the effects of switching to Bazedoxifene 20mg in comparison with switching to calcium 500mg and 400 IU vitamin D (OSTINE) daily on BMD at the femoral neck
BMD at total hip | 6 and 12 months from baseline
  To evaluate the effects of switching to Bazedoxifene 20mg in comparison with switching to calcium 500mg and 400 IU vitamin D (OSTINE) daily on BMD at total hip
Mammography | 12 months from baseline
  Changes in Mammography at12 months from baseline in the Breast Imaging Report and Database System (BI-RADS) classification

OTHER OUTCOMES:
Subject reported treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM) and gastrointestinal symptoms using the Gastrointestinal Symptoms Rating Scale (GSRS)the Spanish versions | At baseline, months 6 and 12
  To evaluate the effects of switching to Bazedoxifene 20mg in comparison with switching to calcium 500mg and 400 IU vitamin D (OSTINE)daily on Subject reported treatment satisfaction using the Treatment Satisfaction Questionnaire for Medication (TSQM) and gastrointestinal symptoms using the Gastrointestinal Symptoms Rating Scale (GSRS)the Spanish versions

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Palacios, MD, Principal Investigator
Locations (3):
- Spain (3):
  - Gabinete Médico Velázquez, Madrid, Madrid
  - Instituto Palacios, Madrid, Madrid
  - Instituto de Ginecología EGR, Madrid, Madrid